CLINICAL TRIAL: NCT03395301
Title: Coil Hysteroscopic Tubal Occlusion : the Treatment of Hydrosalpinx Before IVF-ET
Brief Title: Coil Hysteroscopic Tubal Occlusion in the Treatment of Hydrosalpinx
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Feng Lin, Associate Chief Physician, First Affiliated Hospital of Wenzhou Medical University
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Platinum coils
Record Dates: First submitted 2016-05-19; First posted 2018-01-10 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2017-12

CONDITIONS: Hydrosalpinx
Keywords: hysteroscopy; fiber platinum coil; tubal occlusion

STUDY DESIGN:
Intervention Model Description: Platinum coils were inserted into the tubes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- tubal occlusion (Experimental): Fiber coils were inserted into the interstitial part of fallopian tubes, and IVF-ET was taken out in the following.
  Interventions: Device: Coil

INTERVENTIONS:
Device: Coil — Fiber platinum coil were inserted into the interstitial part of the tubes of patients in hydrosalpinx through hysteroscopy

SUMMARY:
this study is to investigate the success rate of proximal tubal occlusion with coil devices in women with hydrosalinx and to observe there pregnancy rate with IVF-ET.

DETAILED DESCRIPTION:
In this study, investigators will recruit 80 females with unilateral or bilateral hydrosalpinx as confirmed by HSG. Tubal ligation may be a safe and effective method in the treatment of hydrosalpinx. But in this study, investigators will use fiber platinum coils to occlude the tubes. After the treatment, IVF-ET will be applied,and then the patients' pregnancy rate will be assessed in the following-up.

ELIGIBILITY:
Inclusion Criteria:

1. Have unilateral or bilateral hydrosalpinxs as evidenced by HSG.
2. laparoscopic surgery was considered to be contraindicated because of ex-tensive pelvic adhesions.
3. Are willing to undergo a hysterosalpingogram (HSG) 1 months after fiber platinum coil placement to confirm proximal tubal occlusion.
4. Are willing to participate in this clinical study .Are able to comprehend and give informed consent for participation in this study.
5. Have read, understood and signed an informed consent form .

Exclusion Criteria:

1. Active or recent upper or lower pelvic infection
2. Known hypersensitivity to nickel as confirmed by skin test
3. Known allergy to contrast media Pregnancy or suspected pregnancy
4. Evidence of intrauterine abnormalities such as submucous fibroids, polyps, intrauterine adhesions or presence of a uterine septum
5. Poor general or gynecologic health
6. Inability or refusal to provide informed consent

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-30 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 2 months after IVF-ET
  Patients will be followed up with the pregnancy outcomes after the tubal occlusion

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, Gynecologist, Principal Investigator — the 1st affiliated hospital of Wenzhou Medical College
Locations (1):
- the 1st Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matorras R, Rabanal A, Prieto B, Diez S, Brouard I, Mendoza R, Exposito A. Hysteroscopic hydrosalpinx occlusion with Essure device in IVF patients when salpingectomy or laparoscopy is contraindicated. Eur J Obstet Gynecol Reprod Biol. 2013 Jul;169(1):54-9. doi: 10.1016/j.ejogrb.2013.02.008. Epub 2013 Apr 2. PMID 23561020
- [Derived] Wu YC, Huang XF, Yang HY, Chen X, Wang PY, Hu Y, Lin F. Fibered platinum coil: A novel option for the patients of hydrosalpinx with laparoscopic contradiction. Eur J Obstet Gynecol Reprod Biol. 2018 Oct;229:179-184. doi: 10.1016/j.ejogrb.2018.08.579. Epub 2018 Aug 27. PMID 30205314

DOCUMENTS (2):
  • Study Protocol (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03395301/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-01): https://cdn.clinicaltrials.gov/large-docs/01/NCT03395301/SAP_001.pdf